CLINICAL TRIAL: NCT04582825
Title: STROKE-CARD REGISTRY: Extension of Standard Care in Patients With Ischemic Stroke and Transient Ischemic Attack
Brief Title: Stroke-Card Registry
Status: Recruiting | Type: Observational
Sponsor: VASCage GmbH (Other)
Collaborators: Medical University Innsbruck (Other); St John of God Hospital, Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: VASC-E3-2020-04
Record Dates: First submitted 2020-10-03; First posted 2020-10-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Transient Ischemic Attack
Keywords: Stroke secondary prevention; Stroke Risk factors; Biobank; Post-stroke care; Registry
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — Samples will be collected at baseline and the follow-up visits in the department. In addition to plasma (5 aliquots á 500 µL-1000 µL) and serum (5 aliquots á 500 µL per evaluation), a whole blood sample (2.7 mL) will be archived.
  Additionally samples of thrombi extracted by mechanical thrombectomy procedures will be collected for further projects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: N/A - Observational Study — N/A - Observational Study

SUMMARY:
Stroke is the second leading cause of death and one of the main contributors to disability. Patients who survive the acute phase of ischemic stroke and those with transient ischemic attack (TIA) are at high risk of subsequent vascular events. Importantly, recurrent strokes are associated with a higher social and economic impact, higher case fatality, and worse clinical outcome than first-ever strokes. The burden of post-stroke complications, residual deficits, and inadequate medical and psychosocial care all contribute to long-term disability and reduced quality of life in these patients. The Department of Neurology of the Medical University Innsbruck undertook the STROKE-CARD trial (NCT02156778) between 2014 and 2018 with follow-up until 2019 to evaluate the efficacy of the Post-Stroke disease-management program STROKE-CARD care. After implementation of STROKE-CARD care, the investigators aim to document the quality of post-stroke care and compare outcome parameters to historical cohorts and the change over time. Furthermore the investigators aim to gain a large data-resource for future research of biomarkers, disease mechanisms, prognosis and imaging mechanisms for R&D.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and one of the main contributors to disability. Patients who survive the acute phase of ischemic stroke and those with a transient ischemic attack (TIA) are at high risk of subsequent stroke. Importantly, recurrent strokes are associated with a higher social and economic impact, higher case fatality, and worse clinical outcome than first-ever strokes. The burden of post-stroke complications, residual deficits, and inadequate medical and psychosocial care all contribute to long-term disability and reduced quality of life in these patients. Furthermore, effects on quality of life and long-term functional independence are particularly under-investigated.

The Department of Neurology of the Medical University Innsbruck undertook the STROKE-CARD trial (NCT02156778) between 2014 and 2018 with follow-up until 2019 to evaluate the efficacy of the Post-Stroke disease management program STROKE-CARD care. The aim is to evaluate this program in a large multicenter cohort and to establish a biobank of stroke and TIA-patients for future research and development projects.

In brief, the pragmatic and easily implementable STROKE-CARD care program reduced cardiovascular risk and improved health-related quality of life and functional outcome in patients with acute ischemic stroke or TIA in a timeframe of 12 months after the index event. To investigate the effects of STROKE-CARD care on a large basis and over a longer period, an evaluation of approximately 5,000 patients is warranted.

Whereas disease management programs typically rely on expert opinion, the STROKE-CARD initiative moved from a purely empirical approach to a highly structured, individualized, and evidence-based procedure with professional outcome analysis. The STROKE-CARD concept will be implemented in clinical practice and can serve as a model for other disease management initiatives.

Acute and short-term management of stroke and TIA has improved tremendously over the past years with substantial advances in acute therapy, implementation of comprehensive pathways for stroke and TIA, and approval of novel highly effective preventive treatments. As a main unmet challenge in stroke medicine, strategies of long-term care have to be developed and rigorously tested in order to maintain improved short-term patient outcome in the long run.

STROKE-CARD care reduced the one-year cumulative absolute risk of CVD and ameliorated the patients' health-related quality of life at 12 months (EQ-5D-3L overall utility score, P<0.001). These findings were consistent in subgroups according to age, sex, and index event and were robust in the per-protocol analysis. Among pre-specified secondary outcomes assessed at 12 months, the investigators observed improvements in all individual dimensions of the EQ-5D-3L and in one-year functional outcome, that each met the multiplicity-adjusted threshold for statistical significance. Only a few previous trials of disease management programs in stroke and TIA patients have focused on recurrent CVD or quality of life as primary or secondary endpoints and none has considered long-term functional outcome after one year. The previous trial was limited to a 12-month follow-up in selected individuals and the sustainability of benefits of STROKE-CARD care in a large nationwide cohort over a longer follow-up period remains to be determined.

This study aims to detect post-stroke complications, to estimate the patient's demand for nursing services, and support guideline-compliant secondary prevention with full achievement of target levels, lifestyle modifications, and in-person outcome assessment at 3 and 12 months after the index-event, assessment of functional status (impairment), activity (disability), and participation (handicap and health-related quality of life). Additionally, yearly follow-up telephone interviews for cardiovascular outcome and health parameters will be conducted. In case of clinically indicated in-person follow-ups, the interviews will be done in person during the clinical visits. After the implementation of STROKE-CARD care, the investigators aim to document the quality of post-stroke care and compare outcome parameters to historical cohorts and the change over time. Furthermore, the investigators aim to gain a large data resource for future research of biomarkers, disease mechanisms, prognosis and imaging mechanisms for R&D.

The main objective is to evaluate the Post-Stroke Disease Management program STROKE-CARD in a large multicenter cohort of stroke and TIA-patients and to establish a large clinical well-defined cohort. Furthermore, the investigators aim to gain a large data resource for future research of biomarkers, disease mechanisms, prognosis and imaging mechanisms for R&D.

To document and monitor the quality of the Post-Stroke Disease Management program in different centers and compare outcomes to the historical cohort, as well as other published data. Furthermore, the investigators aim to constantly improve post-stroke care. This registry can facilitate to monitor and document the effect on the primary and secondary outcomes.

There will be no formal safety endpoints in this study. No experimental procedures will be applied to patients and most of the procedures done are within the clinical routine. Potential side effects of optimal secondary stroke prevention are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke or high-risk TIA (ABCD2-Score ≥ 4 points) treated at the Department of Neurology of each study center within 30 days after onset
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Patients living outside the catchment area of the participating centers
* Patients under law enforcement or within mandatory military service
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke or high-risk TIA (ABCD2-Score ≥ 4 points) in the last 30 days over 18 years of age will be invited to the study at all study centers in the designated departments.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
CVD outcome | 1-7 years
  CVD outcome defined as nonfatal ischemic stroke, nonfatal hemorrhagic stroke, nonfatal myocardial infarction, or vascular death between hospital discharge and one year in an in-person follow-up and yearly for up to 6 years.
Health-related quality of life: scale | 1-7 years
  Self-reported health-related quality of life after one year in an in-person follow-up and yearly for up to 6 years using a telephone-based follow-up quantified with the European Quality of Life 5-Dimensions 3-Levels (EQ-5D-3L) overall health utility score14 with rescaled European visual analogue scale weights.

SECONDARY OUTCOMES:
Composite stroke event outcome | 1-7 years
  Composite outcome of ischemic stroke, hemorrhagic stroke, or transient ischemic attack (TIA) (defined as transient neurological deficit <24h and absence of diffusion-weighted imaging (DWI) positive lesions on MRI) after one year and on the long run
All-cause mortality | 1-7 years
  All-cause mortality after one year and in the long run
Individual 3-level components of the European Quality of Life 5-Dimensions 3-Levels (EQ-5D-3L) questionnaire | 1-7 years
  Mobility, self-care, usual activities, no pain or discomfort, no anxiety or depression) comparing people reporting no problems (level 1) with those reporting problems (level 2 and 3) after one year in an in-person follow-up and in the long run
Proportions of participants achieving target levels of risk factors | 1-7 years
  * systolic blood pressure <140 mmHg and a diastolic blood pressure <90 mmHg or a systolic blood pressure <130 mmHg and a diastolic blood pressure <85 mmHg at the study visit in patients with diabetes mellitus, severe renal impairment, or small-vessel disease at baseline,
  * achieving a glycated hemoglobin (HbA1c) concentration <7.0% in patients with diabetes mellitus or <8% in selected individuals
  * having quit smoking after one year and on the long run
  * being physically active for an average of >90 minutes/week
  * taking lipid-lowering medication in all patients except those with an event of other determined etiology (e.g. due to vasculitis or vessel dissection)
  * achieving a low-density lipoprotein (LDL) cholesterol concentration <70 mg/dL
  * taking anticoagulation or antiplatelet therapy in patients that had been prescribed such medication
  * taking anticoagulation in patients with atrial fibrillation after one year and in the long run
Functional outcome | 1-7 years
  Good functional outcome defined as modified Rankin Scale25 (mRS) ≤2 after one year and in the long run
  Distribution across mRS categories after one year and in the long run ("shift analysis")

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kiechl, MD, Principal Investigator — Medical University Innsbruck
Locations (2):
- Austria (2):
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Hospital St. John of God, Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toell T, Boehme C, Mayer L, Krebs S, Lang C, Willeit K, Prantl B, Knoflach M, Rumpold G, Schoenherr G, Griesmacher A, Willeit P, Ferrari J, Lang W, Kiechl S, Willeit J. Pragmatic trial of multifaceted intervention (STROKE-CARD care) to reduce cardiovascular risk and improve quality-of-life after ischaemic stroke and transient ischaemic attack -study protocol. BMC Neurol. 2018 Nov 6;18(1):187. doi: 10.1186/s12883-018-1185-2. PMID 30400876
- [Background] Willeit P, Toell T, Boehme C, Krebs S, Mayer L, Lang C, Seekircher L, Tschiderer L, Willeit K, Rumpold G, Schoenherr G, Griesmacher A, Ferrari J, Knoflach M, Lang W, Kiechl S, Willeit J; STROKE-CARD study group. STROKE-CARD care to prevent cardiovascular events and improve quality of life after acute ischaemic stroke or TIA: A randomised clinical trial. EClinicalMedicine. 2020 Jul 28;25:100476. doi: 10.1016/j.eclinm.2020.100476. eCollection 2020 Aug. PMID 32954239
- [Background] Boehme C, Toell T, Mayer-Suess L, Domig L, Pechlaner R, Willeit K, Tschiderer L, Seekircher L, Willeit P, Griesmacher A, Knoflach M, Willeit J, Kiechl S. The dimension of preventable stroke in a large representative patient cohort. Neurology. 2019 Dec 3;93(23):e2121-e2132. doi: 10.1212/WNL.0000000000008573. Epub 2019 Oct 31. PMID 31672716
- [Derived] Karisik A, Dejakum B, Moelgg K, Granna J, Felicetti S, Pechlaner R, Mayer-Suess L, Toell T, Buergi L, Scherer L, Willeit K, Heidinger M, Lang C, Ferrari J, Krebs S, Kleyhons R, Resch H, Willeit J, Seekircher L, Tschiderer L, Willeit P, Sykora M, Schett G, Lang W, Knoflach M, Kiechl S, Boehme C. Incidence, characteristics, and consequences of fractures after acute ischemic stroke and TIA-A prospective cohort study. Int J Stroke. 2025 Oct;20(9):1141-1149. doi: 10.1177/17474930251345300. Epub 2025 May 20. PMID 40391684
- [Derived] Moelgg K, Karisik A, Dejakum B, Felicetti S, Boehme C, Mayer-Suess L, Toell T, Knoflach M, Kiechl S, Pechlaner R. Longitudinal dynamics of pulse wave velocity in the days after acute ischaemic stroke: prospective cohort study. BMJ Open. 2025 Apr 3;15(4):e089304. doi: 10.1136/bmjopen-2024-089304. PMID 40180369
- [Derived] Karisik A, Bader V, Moelgg K, Buergi L, Dejakum B, Komarek S, Eller MT, Toell T, Mayer-Suess L, Pechlaner R, Granna J, Sollereder S, Rossi S, Schoenherr G, Willeit J, Willeit P, Lang W, Kiechl S, Knoflach M, Boehme C; STROKE-CARD study group. Comorbidities associated with dysphagia after acute ischemic stroke. BMC Neurol. 2024 Sep 28;24(1):358. doi: 10.1186/s12883-024-03863-1. PMID 39342159
- [Derived] Komarek S, Dejakum B, Moelgg K, Boehme C, Karisik A, Toell T, Kiechl S, Knoflach M, Pechlaner R, Mayer-Suess L. No association between SARS-CoV-2 vaccination and ischaemic stroke or high-risk transient ischaemic attack. J Neurol Sci. 2024 Jan 15;456:120834. doi: 10.1016/j.jns.2023.120834. Epub 2023 Oct 11. PMID 38134562